CLINICAL TRIAL: NCT03228407
Title: Confocal Endomicroscopy for Permeability of Esophageal Wall in Refractory Gastroesophageal Reflux Disease (GERD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGuire Research Institute (Other)
Collaborators: Hunter Holmes McGuire VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2282
Record Dates: First submitted 2017-07-06; First posted 2017-07-24 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Gastro Esophageal Reflux; Barrett Esophagus; Erosive Esophagitis
MeSH Terms: conditions — Gastroesophageal Reflux; Barrett Esophagus | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigator in the lab performing Ussing's chamber analysis will be blinded to the diagnosis of the patient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Non-erosive reflux disease (NERD) (Active Comparator): Patient's with GERD refractory to PPI with no evidence of erosive esophagitis on endoscopy. Confocal endomicroscopy, endoscopic biopsies and mucosal impedance (MI) will be performed.
  Interventions: Procedure: Confocal endomicroscopy; Diagnostic Test: Endoscopic biopsies; Diagnostic Test: Mucosal impedance (MI)
- Barrett's esophagus/erosive esophagitis (Active Comparator): Patient's with Barrett's esophagus or with erosive esophagitis on endoscopy. Confocal endomicroscopy, endoscopic biopsies and mucosal impedance (MI) will be performed.
  Interventions: Procedure: Confocal endomicroscopy; Diagnostic Test: Endoscopic biopsies; Diagnostic Test: Mucosal impedance (MI)
- Control (Placebo Comparator): Patient's with no h/o GERD or Barrett's esophagus who are undergoing endoscopy for non-GERD related indication. Confocal endomicroscopy, endoscopic biopsies and mucosal impedance (MI) will be performed.
  Interventions: Procedure: Confocal endomicroscopy; Diagnostic Test: Endoscopic biopsies; Diagnostic Test: Mucosal impedance (MI)

INTERVENTIONS:
Procedure: Confocal endomicroscopy — Confocal laser endomicroscopy (CLE) permits real-time in-vivo histologic analysis of esophageal mucosa at the time of upper endoscopy. The technology is based on the principle of illuminating a tissue with a low-power laser and then detecting fluorescent light reflected from the tissue. Because CLE relies upon tissue fluorescence, intravenous fluorescein is generally used to highlight the vasculature and intercellular spaces of the tissue being examined.
  Other Names: cellvizio
Diagnostic Test: Endoscopic biopsies — Additional biopsies will be obtained of the esophageal mucosa.These will be obtained with a standard biopsy forceps inserted through the channel in gastroscope.
Diagnostic Test: Mucosal impedance (MI) — MI balloon measures epithelial impedance along a 10 cm length of esophagus. The gastroscope will be withdrawn and the MI balloon will be advanced into the esophagus through the mouth. The balloon will be inflated so that the sensors contact the esophageal mucosa. After MI measurements are obtained, the balloon will be deflated and withdrawn.

SUMMARY:
Confocal Endomicroscopy for Permeability of Esophageal Wall in Refractory Gastroesophageal Reflux Disease (GERD)

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Ability to give informed consent

Exclusion Criteria:

1. Pregnancy
2. Esophageal varices
3. Prior esophageal or gastric surgery
4. Active gastrointestinal bleeding
5. Evidence of esophageal malignancy
6. Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-04-28 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Correlation between the time from intravenous injection of fluorescein to visualization of fluorescein on probe based confocal endomicroscopy (pCLE) with esophageal permeability (i.e. - epithelial barrier function). | Through study completion, an average of 1 year.

SECONDARY OUTCOMES:
Compare the time from intravenous injection of fluorescein to visualization of fluorescein on probe based confocal endomicroscopy (pCLE) in patients with Barrett's esophagus and controls | Through study completion, an average of 1 year.
Compare the time from intravenous injection of fluorescein to visualization of fluorescein on probe based confocal endomicroscopy (pCLE) in patients with symptoms of refractory GERD and Barrett's esophagus | Through study completion, an average of 1 year.
Correlation between the Ussing's chamber findings (esophageal permeability) and confocal endomicroscopy findings of patients with symptoms of refractory GERD and Barrett's esophagus | Through study completion, an average of 1 year.
Correlation between the Ussing's chamber findings (esophageal permeability) and confocal endomicroscopy findings of patients with symptoms of refractory GERD and controls | Through study completion, an average of 1 year.
Correlation between the Ussing's chamber findings (esophageal permeability) and Mucosal impedance findings of patients with symptoms of refractory GERD and controls | Through study completion, an average of 1 year.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vaezi MF, Choksi Y. Mucosal Impedance: A New Way To Diagnose Reflux Disease and How It Could Change Your Practice. Am J Gastroenterol. 2017 Jan;112(1):4-7. doi: 10.1038/ajg.2016.513. Epub 2016 Dec 13. No abstract available. PMID 27958288
- [Result] Cui R, Zhou L, Lin S, Xue Y, Duan L, Xia Z, Jin Z, Zhang H, Zhang J, Song Z, Yan X. The feasibility of light microscopic measurements of intercellular spaces in squamous epithelium in the lower-esophagus of GERD patients. Dis Esophagus. 2011 Jan;24(1):1-5. doi: 10.1111/j.1442-2050.2010.01083.x. PMID 20626453
- [Result] Tobey NA, Carson JL, Alkiek RA, Orlando RC. Dilated intercellular spaces: a morphological feature of acid reflux--damaged human esophageal epithelium. Gastroenterology. 1996 Nov;111(5):1200-5. doi: 10.1053/gast.1996.v111.pm8898633.
- [Result] Chu CL, Zhen YB, Lv GP, Li CQ, Li Z, Qi QQ, Gu XM, Yu T, Zhang TG, Zhou CJ, Rui-Ji, Li YQ. Microalterations of esophagus in patients with non-erosive reflux disease: in-vivo diagnosis by confocal laser endomicroscopy and its relationship with gastroesophageal reflux. Am J Gastroenterol. 2012 Jun;107(6):864-74. doi: 10.1038/ajg.2012.44. Epub 2012 Mar 13. PMID 22415199